CLINICAL TRIAL: NCT04821817
Title: The Effect of Rocuronium as an Anesthetic Adjuvant in Peribulbar Anesthesia for Adult Strabismus Surgery: Randomized Controlled Double-blind Study
Brief Title: Peribulbar Rocuronium in Adult Strabismus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Assistant Professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 34506/2/21
Record Dates: First submitted 2021-03-24; First posted 2021-03-30 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Strabismus; Regional Anesthesia Morbidity; Rocuronium
Keywords: Strabismus; peribulbar anesthesia; rocuronium; akinesia
MeSH Terms: conditions — Strabismus | interventions — Saline Solution; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * The patients will be blinded to their groups.
  * An anesthesia resident who will not participate in the study and have no subsequent rule in it will help in the preparation of local anesthetic mixtures under strict aseptic precautions.
  * The anesthetist who will perform the peribulbar block will be blinded to the local anesthetic mixtures he will inject.
  * An assistant nurse who will be blinded to the study groups and will have no subsequent rule in it will help in a collection of the data of measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Control group) (Placebo Comparator): Patients in this group will receive peribulbar anesthesia with 10 ml local anesthetic mixture composed of 4 ml of plain bupivacaine 0.5%, 4 ml of lidocaine 2% containing 50 IU, and 2 ml normal saline.
  Interventions: Drug: Normal saline
- Group R (rocuronium group) (Experimental): Patients in this group will receive peribulbar anesthesia with 10 ml local anesthetic mixture composed of 4 ml of plain bupivacaine 0.5%, 4 ml of lidocaine 2% containing 50 IU, and 0.06 mg/kg of rocuronium in 2 ml normal saline.
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Normal saline — peribulbar anesthesia with 10 ml local anesthetic mixture composed of 4 ml of plain bupivacaine 0.5%, 4 ml of lidocaine 2% containing 50 IU, and 2 ml normal saline.
  Arms: Group C (Control group)
Drug: Rocuronium — peribulbar anesthesia with 10 ml local anesthetic mixture composed of 4 ml of plain bupivacaine 0.5%, 4 ml of lidocaine 2% containing 50 IU, and 0.06 mg/kg of rocuronium in 2 ml normal saline.
  Arms: Group R (rocuronium group)

SUMMARY:
* This is a prospective randomized clinical study that will be carried on adult patients aged from 21-60 years and presented for strabismus surgery under peribulbar anesthesia.
* Patients will be excluded if they refused to participate or had a contraindication to peribulbar anesthesia.
* Patients will be randomly distributed into either control group in which peribulbar anesthesia will be performed by injection of 10 ml local anesthetic mixture composed of 4 ml of plain bupivacaine 0.5%, 4 ml of lidocaine 2% containing 50 IU, and 2 ml normal saline or rocuronium group which peribulbar anesthesia will be performed by injection of 10 ml local anesthetic mixture composed of 4 ml of plain bupivacaine 0.5%, 4 ml of lidocaine 2% containing 50 IU, and 0.06 mg/kg of rocuronium in 2 ml normal saline.
* Measurements will include; -

  1. Patient age, weight, height, gestational age, and gravidity.
  2. The duration of globe akinesia (primary outcome).
  3. The onset of lid and globe akinesia and the duration of lid akinesia
  4. The onset and duration of sensory block
  5. Time required to start the surgery
  6. Akinesia score
  7. The visual analog score (VAS) which is composed of 0-10 score will be used to assess the severity of postoperative pain (where 0=no pain and 10=severe pain), The VAS score will be evaluated 1 h, 2 h postoperative, then every 2 h till 12 h. Any patients with VAS score more than 4 received rescue analgesia in the form of 50 mg tramadol intravenous injection with the calculation of the time for the first call of postoperative analgesia.
  8. Any detected complication as nausea and vomiting, pain on injection, or increased intraocular tension.

DETAILED DESCRIPTION:
This prospective randomized double-blind study will be carried out on adult patients who will be presented for strabismus surgery in Ophthalmology Department in Tanta university hospitals over the 6-month duration, an informed written consent will be obtained from all the participants, all patients data will be confidential and will be used for the current study only.

The patients will be randomly allocated into two groups with the aid of computer-generated software of randomization. All the local anesthetic mixtures will be prepared under complete aseptic precautions by an anesthesia resident who will not participate in the study and will be blinded to its groups in to: - Group C (Control group) (20 Patients): Patients in this group will receive peribulbar anesthesia with a 10 ml local anesthetic mixture composed of 4 ml of plain bupivacaine 0.5%, 4 ml of lidocaine 2% containing 50 IU, and 2 ml normal saline.

Group R (rocuronium group) (20 patients): Patients in this group will receive peribulbar anesthesia with 10 ml local anesthetic mixture composed of 4 ml of plain bupivacaine 0.5%, 4 ml of lidocaine 2% containing 50 IU, and 0.06 mg/kg of rocuronium in 2 ml normal saline.

Anesthetic technique On arrival of patients to the pre-anesthesia preparation room, we will allow them to rest in a supine position with the connection of monitors that consist of 5 leads ECG, non-invasive blood pressure, pulse oximeter, and temperature. Also, intravascular access will be obtained.

Once the patient will be admitted to the operating theatre, all monitors will be applied. A nasal cannula was used at a flow rate of 2-4 l/min to supply oxygen to patients. The peribulbar block will be performed by the same anesthesiologist under aseptic precautions.

The technique of peribulbar block Disposable needles in a size of 25 gauge and 16mm bevels will be used to perform the peribulbar injection. The injection site will be limited by the lateral nasal margin laterally, inferior orbital margin inferiorly, and the lower lacrimal punctum superiorly. Once the needle introduced, the patient will be asked to look in the four cardinal directions of the gaze, superior, inferior, nasal, and temporal to ensure that the needle is not penetrating the eye globe, then negative aspiration will be done to exclude intravascular position of the needle, then, the peribulbar injection of the previously prepared local anesthetic mixture will be performed over 30 seconds and followed by the fullness of the eyelids.

The eyelids will be closed and covered by eye pads carefully with an application of 20 mmHg pressure through an intermittent application of Honan ball for 10 min. The intermittent eye compression will be relieved after 1 min, 3 min, 5 min, 7 min, 9 min, and 10 min to assess the onset and the quality of sensory and motor blockade. The sensory block will be assessed by the abolishment of corneal reflex to the installation of physiological drops on the cornea or conjunctiva. The onset of anesthesia will be determined by the time interval from local anesthetics injection and loss of corneal reflex. The motor block will be evaluated by asking the patient to open, close, and squeeze his eye (Lid Akinesia) and to move his eye globe in the four directions of the gaze (globe akinesia). The quality of akinesia will be assessed through the use of akinesia score where 0=inability to move (total akinesia), 1=partial movement (partial akinesia), and 2=full movements (no akinesia). This score was used to assess both lid akinesia and globe akinesia in the four directions with an overall score of 10.

The onset of lid akinesia will be calculated from peribulbar injection to the partial loss of ability to open or squeeze eyelids, while the onset of globe akinesia will be estimated from the injection of the local anesthetic mixture and partial loss of movement of the eye globe in the four cardinal directions. The surgery will be considered to be optimal to be started when the patient had corneal anesthesia together with partial lid and globe akinesia. The optimal time to start the surgery will be considered as the elapsed time between local anesthetics injection and satisfying the goals to start the surgery. The intraocular pressure will be measured preoperatively and immediately before initiating the surgery with detection of a number of patients with an increase in the intraocular tension (increase intraocular pressure more than 25 mmHg or by more than 10 mmHg than the preoperative value).

The duration of the sensory block will be estimated to be the time interval from the peribulbar injection till regaining corneal sensation, while, the duration of lid or globe akinesia will be determined by the time elapsed between performing the peribulbar injection and the full regaining of lid or globe movement respectively.

The primary outcome will be the duration of globe akinesia. Secondary outcomes will include the onset and duration of sensory block.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Aged 21- 60 years
* American Society of Anesthesiologists class (ASA) I to III
* presented for elective strabismus surgery under peribulbar anesthesia.

Exclusion Criteria:

* Patient refusal to participate.
* uncooperative patient.
* Neurological disorders.
* Psychological disorders
* Suspected or diagnosed coagulopathy.
* Known allergy to the used medications.
* Ocular infection
* Co-existing glaucoma

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-04-03 (Actual); Primary Completion 2025-02-09 (Actual); Study Completion 2025-02-09 (Actual)

PRIMARY OUTCOMES:
The duration of globe akinesia | up to first 2 hours intraoperative
  Time interval from reaching the highest lid and globe akinesia score till restoration of the full lid and globe movement

SECONDARY OUTCOMES:
The onset of sensory block | Intraoperative (every 2 minutes after peribulbar injection)
  Time interval from peribulbar injection till loss of corneal sensation
The duration of sensory block | Intraoperative (Every 30 minutes in the first 4 hours)
  time interval from the peribulbar injection till regaining corneal sensation,

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Abdelkhalik, M.D, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Algharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data of primary outcome will be available with the corresponding author till 6 months after approval of the publication of the trial.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after approval of the publication of the trial.
Access Criteria: Contact the principle investigator